CLINICAL TRIAL: NCT02405962
Title: Effects of a Parental Training Program Using Group-based Acceptance and Commitment Therapy for Managing Children With Asthma: a Randomized Controlled Trial
Brief Title: Training Parents by Acceptance and Commitment Therapy for Managing Childhood Asthma Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Yim Wah MAK, Ph.D, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20150109001
Record Dates: First submitted 2015-03-28; First posted 2015-04-01 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Childhood Asthma
Keywords: Acceptance and Commitment Therapy; Childhood asthma; Randomized controlled trial; Training parents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Parents of children with asthma will receive one session of asthma educational talk as the usual care, plus three weekly sessions of telephone calls to assess the child's asthma symptoms
  Interventions: Behavioral: Control
- ACT group (Experimental): Parents of children with asthma will receive four sessions of group-based ACT intervention integrated with asthma education (its content will be the same as that of the Control Group).
  Interventions: Behavioral: ACT

INTERVENTIONS:
Behavioral: ACT — Four sessions of group-based ACT integrated with asthma education. Each session will compose of pediatric asthma education based on guidelines of Global Strategy for Asthma Management and Prevention Revised 2011, plus group-based Acceptance and Commitment Therapy (ACT). The goal of ACT is to enhance the psychological flexibility of the parents, enabling them to (1) become aware of their thoughts and feelings regarding their child's asthma and its management, (2) accept and adapt flexibly to challenging situations, and (3) take actions to achieve valued goals in childhood asthma management.
  Arms: ACT group
Behavioral: Control — One session of educational talk about pediatric asthma care, as the usual care. To ensure the equivalency of the assigned sessions between groups, after attending the talk in the first week, the parents in the Control group will receive three telephone calls, starting from the second week on a weekly basis. This arrangement can also minimize the interference of the usual care naturalistically available in the study setting.
  Arms: Control group

SUMMARY:
The purpose of this study is to examine whether a parental training program using group-based Acceptance and Commitment Therapy for childhood asthma care, is effective in reducing the children's unplanned health care services utilization and asthmatic symptoms.

DETAILED DESCRIPTION:
One-tenth of children in worldwide are diagnosed with asthma and it is the leading cause for unplanned health care services utilization. Parents, as the primary caregivers, experience different level of psychological distress in taking care of their children with asthma. Some of them responded with avoidance-based coping, which results in poor asthma symptom management and monitoring. Acceptance and Commitment Therapy (ACT) is a contextual focused, behavioral therapy aiming at improving psychological flexibility, so that a person can be more opened up to engaging in value-driven behavior modification, thus attaining an optimal disease control. The benefits of ACT have been demonstrated on both parents and their children with chronic health conditions such as developmental disabilities, acquired brain injuries, chronic pain, cancer and mental disorders. To date, no ACT intervention has been conducted on examining its effects on training parents in managing their children with asthmatic conditions.

This is the first study aims to examine the effects of a parental training program using group-based Acceptance and Commitment Therapy (ACT) in reducing the unplanned health care services utilization and asthmatic symptoms, among children with asthma. Parents of children diagnosed with asthma will either receive one session of pediatric asthma educational talk as usual practice in the study hospital, or in addition, four sessions of group-based ACT integrated with asthma education.

If the group-based ACT is effective in reducing children's asthmatic symptoms and overall unplanned asthma-related health services utilization, it could lead to substantial health benefits in children with asthma and on parents with a reduction in psychological distress. In addition to cutting medical expenses, it could also contribute to the community health through the reduction in mortality and morbidity due to asthmatic attacks. Furthermore, information collected from this proposed study will open up an opportunity for exploring the potential of ACT-based intervention in managing other childhood chronic diseases.

ELIGIBILITY:
Inclusion Criteria for parents:

* Between 18 and 65 years old
* Fathers or mothers in each family who are primarily responsible for the daily care of their child with asthma
* Living together with the index child
* Able to communicate in Cantonese
* Hong Kong residents who plan to stay in Hong Kong for at least 6 months
* Accessible by telephone and by mail

Inclusion Criteria for children:

* 3 to 12 years old with a physician's diagnosis of asthma

Exclusion criteria for parents:

* Enrolled in another asthma research intervention study

Exclusion criteria for children:

* Enrolled in another asthma research intervention study
* Two years old or under presented with an acute wheezing attack. As symptoms at this age can be due to bronchiolitis, a viral infection, rather than asthma
* Have (1) other chronic pulmonary diseases, such as cystic fibrosis (CF), bronchopulmonary dysplasia (BPD), oxygen dependent conditions, or presence of tracheotomy; (2) other significant medical and mental morbidities, such as congenital malformation, Down's syndrome, cerebral palsy and psychomotor retardation. Both may hinder the control of asthma.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yim Wah Mak, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (3):
- Hong Kong (3):
  - School of Nursing, The Hong Kong Polytechnic University, Hung Hom, Kowloon
  - Ambulatory Care Clinic, Department of Paediatrics and Adolescent Medicine, Tuen Mun Hospital, Hong Kong
  - Pediatric asthma nurse-led clinic, Department of Paediatrics and Adolescent Medicine, Tuen Mun Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chong YY, Mak YW, Leung SP, Lam SY, Loke AY. Acceptance and Commitment Therapy for Parental Management of Childhood Asthma: An RCT. Pediatrics. 2019 Feb;143(2):e20181723. doi: 10.1542/peds.2018-1723. Epub 2019 Jan 18. PMID 30659063

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled parents of children aged 3-12 years who had been diagnosed with asthma from 2 pediatric respiratory outpatient clinics, the Ambulatory Care Centre and a nurse-led asthma clinic, in the Department of Pediatrics and Adolescent Medicine of a public hospital under the Hospital Authority in Hong Kong.
Pre-assignment Details: No significant events in this study occurred after participant enrollment. All the enrolled participants who provided written consent to participate in the study were included in the study.
Groups:
- Control Group: Parents of children with asthma will receive one session of asthma educational talk as the usual care, plus three weekly sessions of telephone calls to assess the child's asthma symptoms
  Control: One session of educational talk about pediatric asthma care, as the usual care.
  To ensure the equivalency of the assigned sessions between groups, after attending the talk in the first week, the parents in the Control group will receive three telephone calls, starting from the second week on a weekly basis. This arrangement can also minimize the interference of the usual care naturalistically available in the study setting.
Period: Overall Study
Arm/Group | Control Group | ACT Group
Started | 84 | 84
Post-intervention | 80 | 81
3 Months After the Intervention | 80 | 79
Completed | 83 | 79
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 4
Not completed — A participant has moved to another place | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | ACT Group | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.07 (6.19) | 37.74 (5.55) | 38.40 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 76 | 148
  Male | 12 | 8 | 20
Region of Enrollment [Number; unit: participants]
  Hong Kong | 84 | 84 | 168
Educational attainment [Count of Participants; unit: Participants]
  Primary education or below | 5 | 4 | 9
  Secondary education | 65 | 58 | 123
  Tertiary education or above | 14 | 22 | 36
Monthly household income (Hong Kong Dollars) [Count of Participants; unit: Participants]
  < $ 10,000 | 15 | 10 | 25
  $10,000 to $25,000 | 27 | 18 | 45
  $25,001 to $50,000 | 37 | 51 | 88
  >$50,000 | 5 | 5 | 10
Employment status [Count of Participants; unit: Participants]
  Full-time employed | 34 | 29 | 63
  Part-time employed | 6 | 6 | 12
  Home-makers or unemployed | 44 | 49 | 93
Marital status [Count of Participants; unit: Participants]
  Single/ separated/ divorced/ widowed | 12 | 11 | 23
  Married | 72 | 73 | 145
Smoking status [Count of Participants; unit: Participants]
  Both parents are non-smokers | 53 | 51 | 104
  At least one parent is a current smoker | 31 | 33 | 64
History of asthma diagnosis [Count of Participants; unit: Participants]
  Neither parents has a history of asthma | 48 | 51 | 99
  At least one parent has a history of asthma | 24 | 22 | 46
  Other family members has a history of asthma | 12 | 11 | 23
Child's age [Mean (Standard Deviation); unit: years] | 6.95 (2.46) | 6.67 (2.55) | 6.81 (2.50)
Child's gender [Count of Participants; unit: Participants]
  Male | 52 | 51 | 103
  Female | 32 | 33 | 65
Child's age of diagnosis as asthma [Mean (Standard Deviation); unit: years] | 3.61 (1.88) | 3.31 (1.70) | 3.46 (1.79)
Child's concurrently diagnosed with allergic rhinitis [Count of Participants; unit: Participants]
  Yes | 30 | 29 | 59
  No | 54 | 55 | 109
Child's concurrently diagnosed with eczema [Count of Participants; unit: Participants]
  Yes | 8 | 10 | 18
  No | 76 | 74 | 150
Child's current use of oral Montelukast as prophylaxis [Count of Participants; unit: Participants]
  Yes | 13 | 11 | 24
  No | 71 | 73 | 144
Child's current use of inhaled corticosteroid as prophylaxis, by types [Count of Participants; unit: Participants]
  None | 33 | 47 | 80
  Beclometasone dipropionate | 46 | 35 | 81
  Fluticasone propionate | 4 | 1 | 5
  Fluticasone propionate and Salmeterol | 1 | 1 | 2
Child use 1 or more course of oral prednisolone use in the previous year due to asthma exacerbations [Count of Participants; unit: Participants]
  Yes | 44 | 50 | 94
  No | 40 | 34 | 74
Child's total number of GOPC visits due to asthma exacerbations in the past 6 months [Count of Participants; unit: Participants] — This measure refers to the total number of GOPC (general outpatient clinic) visits due to asthma exacerbations in the past 6 months
  Participants
    0 times | 74 | 69 | 143
    1 to 2 times | 5 | 10 | 15
    3 to 4 times | 4 | 3 | 7
    5 times or above | 1 | 2 | 3
Child's total number of PP clinic visits due to asthma exacerbations in the past 6 months [Count of Participants; unit: Participants] — This measure refers to the child's total number of PP private practitioners' clinic visits due to asthma exacerbations in the past 6 months
  Participants
    0 times | 46 | 47 | 93
    1 to 2 times | 26 | 22 | 48
    3 to 4 times | 9 | 7 | 16
    5 times or above | 3 | 8 | 11
Child's total number of emergency care visit(s) due to asthma exacerbations in the past 6 months [Count of Participants; unit: Participants]
  0 times | 54 | 49 | 103
  1 to 2 times | 26 | 29 | 55
  3 to 4 times | 3 | 5 | 8
  5 times or above | 1 | 1 | 2
Child's total number of hospital admission(s) due to asthma exacerbation(s) in the past 6 months [Count of Participants; unit: Participants]
  0 times | 67 | 60 | 127
  1 to 2 times | 16 | 22 | 38
  3 to 4 times | 1 | 2 | 3
Child's use of alternative therapy in the past 6 months, by types [Count of Participants; unit: Participants]
  None | 73 | 74 | 147
  Herbal soup | 9 | 8 | 17
  Natural moxibustion | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Child's Total Number of Emergency Department Visits Due to Asthma Attacks Over the 6 Months Post Intervention
Description: Parental report of the total number of emergency department visits due to asthma attacks of a child in either a / public hospital(s) of the Hong Kong Hospital Authority and/or a private hospital(s) over 6 months post intervention
Time Frame: 6 months after the completion of intervention
Measure: Mean (Standard Error); unit: Number of visits
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of visits | 0.38 (0.11) | 0.08 (0.04)
Statistical Analysis 1: Comparison: Control Group vs ACT Group; Test type: Superiority; p < 0.05, Mixed Models Analysis; Adjusted Incidence Rate Ratio = 0.20, 95% CI 2-sided [0.08 to 0.53]

2. Secondary Outcome: Children's Total Number of General Outpatient Clinic Visits Due to Asthma Attacks Over the Past 6 Months
Description: The total number of general outpatient clinic visits due to asthma attacks of children over the past 6 months by parental reports in self-administered questionnaires
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of visits
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of visits | 0.18 (0.06) | 0.05 (0.02)

3. Secondary Outcome: Children's Total Number of Private Practitioner's Clinic Visits Due to Asthma Attacks Over the Past 6 Months
Description: The total number of private practitioner's clinic visits due to asthma attacks of children over the past 6 months by parental reports in self-administered questionnaires
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of visits
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of visits | 0.85 (0.14) | 0.40 (0.09)

4. Secondary Outcome: Children's Total Number of Hospital Admissions Due to Asthma Attacks Over the Past 6 Months
Description: The total number of hospital admissions due to asthma attacks of children in either the public hospitals under the Hong Kong Hospital Authority and/or the private hospitals over the past 6 months by parental reports in self-administered questionnaires
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of hospital admissions
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of hospital admissions | 0.06 (0.03) | 0.04 (0.02)

5. Secondary Outcome: Children's Number of Days of Hospital Stay Due to Asthma Attacks Over the Past 6 Months
Description: The total number of days of inpatient hospital stay due to asthma attacks of children in either the public hospitals under the Hong Kong Hospital Authority and/or the private hospitals over the past 6 months by parental reports in self-administered questionnaires
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of days of hospital stay
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of days of hospital stay | 3.75 (0.42) | 3.67 (0.72)

6. Secondary Outcome: Children's Asthma Symptoms During Daytime Per Week Over the Past 4 Weeks
Description: The days per week that the child presented with asthma symptoms (either chronic coughing, wheezing, shortness of breath, or chest tightness) during the daytime over the past 4 weeks, assessed by parental reports in self-administered questionnaires
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of days
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of days | 2.30 (0.22) | 0.58 (0.15)

7. Secondary Outcome: Children's Asthma Symptoms During Nighttime Per Week Over the Past 4 Weeks
Description: The nights per week that the child was awakened due to asthma symptoms (either chronic coughing, wheezing, shortness of breath, or chest tightness) during the nighttime over the past 4 weeks, assessed by parental reports in self-administered questionnaires
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of nights
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of nights | 1.89 (0.23) | 0.55 (0.13)

8. Secondary Outcome: Children's Days of Activities Affected by Asthma Symptoms Per Week Over the Past 4 Weeks
Description: The days per week that the child has to slow down or discontinue his/her activities due to asthma symptoms (either chronic coughing, wheezing, shortness of breath, or chest tightness) over the past 4 weeks, assessed by parental reports in self-administered questionnaires.
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of days
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of days | 0.84 (0.16) | 0.17 (0.07)

9. Secondary Outcome: Children's Reliever Use Due to Asthma Symptoms Per Week Over the Past 4 Weeks
Description: The days per week that the child requires to use an inhaled bronchodilator to relieve asthma symptoms (either chronic coughing, wheezing, shortness of breath, or chest tightness) over the past 4 weeks, assessed by parental reports in self-administered questionnaires
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: Number of days
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
Number of days | 1.62 (0.22) | 0.59 (0.15)

10. Secondary Outcome: Parents' Psychological Flexibility
Description: The Acceptance and Action Questionnaire-II was used to assess the psychological flexibility of the parents.
  The parents rated 7 statements on a 7-point Likert scale ranging from 1 (never true) to 7 (always true), for example: "My painful experiences and memories make it difficult for me to live a life that I would value." The possible range of the total score is 7-49 (minimum value = 7; maximum value = 49). A higher score means a worse outcome, that is the parent is more psychologically inflexible.
  The Acceptance and Action Questionnaire-II possessed good internal consistencies (mean Cronbach's alpha (α) = .84, range α = .86 to .88) and test-retest reliabilities over a 3-month interval (test-retest reliability coefficient (r) = .81) and 12-month interval (r = .79), respectively.
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
score on a scale | 20.40 (0.89) | 14.67 (0.72)

11. Secondary Outcome: Parents' Psychological Adjustment to Their Child's Asthma
Description: The Parent Experience of Child Illness scale was used to capture the psychological adjustment of parents in caring for a child with asthma.
  The Parent Experience of Child Illness scale contains 25 statements with 3 subscales for assessing the illness-specific psychological distress experienced by parents who have a chronically ill child, including Guilt and Worry, Unresolved Sorrow and Anger, and Long-term Uncertainty, together with 1 subscale on perceived Emotional Resources. The possible range of each of the subscale score is 0-4 (minimum value = 0; maximum value = 4). Higher scores in Guilt and Worry, Unresolved Sorrow and Anger, and Long-term Uncertainty mean worse outcomes. A higher score in Emotional Resources means a better outcome.
  The Parent Experience of Child Illness scale had adequate internal consistencies (α in each subscale = .72 to .89) and test-retest reliabilities over a 2-week interval (r in each subscale = .83 to .86)
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: score on a subscale
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
score on a subscale
  Guilt and worry | 1.46 (0.07) | 1.19 (0.06)
  Unresolved sorrow and anger | 1.16 (0.07) | 0.95 (0.05)
  Long-term uncertainty | 1.13 (0.08) | 0.98 (0.06)
  Perceived emotional resources | 2.38 (0.10) | 2.64 (0.08)

12. Secondary Outcome: Parents' Psychological Symptoms
Description: The Depression Anxiety Stress Scale 21 was used to evaluate the psychological symptoms of parents.
  This instrument contains 21 statements with 3 subscales assessing the symptoms of depression, anxiety and stress of parents, respectively. The parents rated the degree to which each statement applied to them in the past week on a 4-point Likert scale from 0 (does not apply to me at all) to 3 (applies to me very much, or most of the time).
  The subscale scores for depression, anxiety and stress subscale would be multiplied by two. The possible range for each of the subscale score is 0-42 (minimum value = 0, maximum value = 42). Higher scores mean worse outcomes. The cut-off scores indicating at least a mild level of psychological symptoms of an individual are 9 for depression; 7 for anxiety and 14 for stress, respectively.
  The Cronbach's alpha for the depression, anxiety, and stress subscales in DASS-21 were 0.82, 0.88 and 0.90, respectively.
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: score on a subscale
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
score on a subscale
  Depressive symptoms | 4.12 (0.58) | 2.75 (0.40)
  Anxiety symptoms | 6.10 (0.65) | 3.80 (0.42)
  Stress symptoms | 9.85 (0.90) | 7.41 (0.63)

13. Secondary Outcome: Parents' Knowledge in Childhood Asthma Management
Description: The Asthma Knowledge Questionnaire was used to assess the knowledge level among parents in pediatric asthma management.
  This instrument composes of 25 true and false statements to measure parental asthma knowledge, including symptoms, triggers, treatment and prevention (Cronbach's alpha = 0.69).
  The possible range of total score is 0-25 (minimum value = 0; maximum value = 25). A higher score means a better outcome, that is the parent has better asthma knowledge.
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
score on a scale | 18.81 (0.29) | 19.50 (0.27)

14. Secondary Outcome: Parents' Asthma Management Self-efficacy
Description: The Parental Asthma Management Self-Efficacy Scale was used to assess the self-efficacy of parents in childhood asthma care.
  The instrument consists of 13 questions with two subscales in assessing the self-efficacy of parents in preventing and in managing children's asthma attacks. The parents rated the strength of their beliefs in a variety of situations related to childhood asthma management on a 5-point rating scale from 1 (not at sure) to 5 (completely sure). The possible range of each of the subscale score is 1-5 (minimum value = 1, maximum value = 5). A higher score means a better outcome, that is the parent has better self-efficacy.
  This instrument had satisfactory internal consistency (α of each subscale = .77 to .82) and strong construct validity with the self-efficacy of children in managing asthma (r = 0.36).
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: score on a subscale
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
score on a subscale
  Attack prevention | 3.89 (0.07) | 4.10 (0.07)
  Attack management | 3.59 (0.08) | 3.81 (0.05)

15. Secondary Outcome: Parents' Quality of Life
Description: The Pediatric Asthma Caregiver's Quality of Life was used to assess the quality of life of the parents in caring for a child with asthma.
  This instrument is a 13-question, 7-point Likert scale measuring parental psychosocial well-being with 2 subscales, emotional function and activity limitation. The possible range of each of the subscale score is 1-7 (minimum value = 1, maximum value = 7). Higher scores in the subscales mean better outcomes, that is the parent has a better quality of life.
  This instrument had stable reliabilities within the intervals of four weeks (intraclass correlation coefficient (ICC) = 0.80 to 0.85).
Time Frame: At 6 months after the intervention
Measure: Mean (Standard Error); unit: score on a subscale
Arm/Group | Control Group | ACT Group
Number analyzed (Participants) | 84 | 84
score on a subscale
  Emotional function | 5.36 (0.12) | 5.69 (0.10)
  Activity limitation | 5.23 (0.13) | 5.65 (0.11)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Control Group: Participants will receive one session of educational talk on childhood asthma management (Intervention as usual).
- ACT Group: Participants will receive four sessions of group-based Acceptance and Commitment Therapy integrated with the asthma education that provided to the participants of the control group.
Arm/Group | Control Group | ACT Group
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84
Other Adverse Events (participants affected / at risk) | 0/84 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No